CLINICAL TRIAL: NCT01851837
Title: Response Of Weight And Lipid Profile To Exercise Time In Sedentary Overweight/Obese Middle-Aged And Older Women
Brief Title: Exercise Time in Sedentary Middle-aged Female
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: P.L.Shupik National Medical Academy of Post-Graduate Education (Other)
Responsible Party: Principal Investigator, Mohammadreza Rezaeipour, MD, PhD, Assistant professor, University of Sistan and Baluchestan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: no grant
Record Dates: First submitted 2013-05-04; First posted 2013-05-13 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2016-05

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): Study group I (57 participants) received the continuous training of exercise time.
  Interventions: Other: Exercise time
- Group II (Active Comparator): Study group II (58 participants) received the interval training of exercise time.
  Interventions: Other: Exercise time

INTERVENTIONS:
Other: Exercise time — Continuous training, Interval training

SUMMARY:
The exercise time is an important factor among the medical guides for weight loss; however, there is still little knowledge about exercise duration paths in middle-aged and older women. The present study aimed to determine the effects of the interval training on weight loss and lipid profile, and to compare its efficiency with the continuous training.

DETAILED DESCRIPTION:
Participants included sedentary women (age 45-75 years) with overweight or obesity (n= 115). They were randomly divided into two groups including continuous exercise, and interval exercise. The weight assessment parameters including change in weight and body composition, blood sample tests were performed pre- and three month post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle
* Good Health
* Weight stability

Exclusion Criteria:

*Abnormality or history of Disease

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
HDL-c | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Mohammadreza Rezaeipour, M.D., Principal Investigator — Member of Scientific Board in Physical Education and Sport Sciences